CLINICAL TRIAL: NCT02610504
Title: A 26 Week Prospective Open Label Clinical Study Evaluating A Single Intra-Articular Injection of Durolane 3ml for Treatment of Osteoarthritis Pain of the Shoulder
Brief Title: Prospective Single Center Open Label Study of Shoulder OA Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13DUR503
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis
Keywords: degenerative arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Durolane 3ml (Experimental): Single intra-articular injection into shoulder
  Interventions: Device: Durolane

INTERVENTIONS:
Device: Durolane — single injection of 3ml
  Other Names: Hyaluronic Acid

SUMMARY:
Open label, prospective, single cohort study of Durolane 3ml intra-articular injection into the shoulder for pain in mild to moderate patients

DETAILED DESCRIPTION:
Subjects 19-85 years old will receive a single intra-articular (IA) injection of DUROLANE® 3mL given for the relief of pain in the treatment of symptomatic osteoarthritis (OA) of the shoulder followed over a 26-week time period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glenohumeral osteoarthritis
* SPOM score greater than or equal to 50 in study shoulder
* Willing to discontinue oral and topical analgesia other than rescue acetaminophen
* abstinence from any other IA or per-articular injections for the shoulder during the course of the trial
* patients with chronic shoulder pain lasting more than 6 months without clinically significant improvement in pain over the past one month
* pain at least 50% of the days during previous month
* patients who have failed conventional therapy of NSAIDs or steroid injections
* patients with a retained active range of motion of at least 30% in all directions to rule out frozen shoulder
* cooperative and able to communicate effectively
* agree not to participate in any other studies during trial

Exclusion Criteria:

* significant pain from other joints requiring chronic analgesic therapy
* presence of one or more conditions besides OA that could confound pain and functional assessments
* clinically apparent tense effusion, malalignment or instability in study shoulder
* shoulder x-rays of acute fractures, sever loss of bone density, avascular necrosis or severe deformity
* inability to abstain from analgesic use other than rescue acetaminophen
* IA injections of steroids to the study shoulder within 3 months or any other joint within the prior month
* IA injection of hyaluronic acid in the study shoulder within 9 months of baseline
* allergic reaction to HA
* any medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion or may compromise pain assessments of shoulder
* uncontrolled hypothyroidism
* pregnant or breastfeeding women
* planned surgical procedure
* history or presence of septic arthritis of study joint or active skin disease or infection in the area of the injection site
* treatment with glucosamine/chondroitin initiated or unstable within 3 months of baseline or change in physical therapy for the study shoulder within 1 month of baseline

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Shoulder pain on movement (SPOM) 0-100mm VAS | over 26 weeks

SECONDARY OUTCOMES:
Shoulder pain at night (SPAN) 0-100mm VAS | over 26 weeks
American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment form | over 26 weeks
Patient Global Assessment (PGA) | over 26 weeks
Shoulder pain rescue medication diary | over 26 weeks
Adverse events, concomitant medications, physical exam | over 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael McKee, MD, Principal Investigator — St. Michaels Hospital
Locations (1):
- St. Michaels Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2015-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT02610504/Prot_000.pdf